CLINICAL TRIAL: NCT04644939
Title: Impact of Telephone Call for Patient Education on Bowel Preparation Quality in Outpatient Colonoscopies
Brief Title: Impact of Telephone Call on Bowel Preparation Quality in Colonoscopies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Dr. Walid Nassreddine, Head of Gastroenterology division, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10112020
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Colonoscopy
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Patients will receive bowel preparation instructions in a conventional way in addition to a telephone call for education purposes one day prior to procedure
  Interventions: Other: Phone calls; Other: Colonoscopy
- Conventional group (Placebo Comparator): Patients will receive bowel preparation instructions in a conventional way
  Interventions: Other: Standard bowel preparation; Other: Colonoscopy

INTERVENTIONS:
Other: Phone calls — Patients undergoing outpatient colonoscopy will receive the standard bowel preparation instructions and a telephone call one day before the procedure to re-explain the instructions and the importance of bowel preparation
  Arms: Interventional group
Other: Standard bowel preparation — Patients undergoing outpatient colonoscopy will receive the standard bowel preparation instructions
  Arms: Conventional group
Other: Colonoscopy — Patients will undergo colonoscopy

SUMMARY:
Bowel preparation regimens typically incorporate dietary modifications along with oral cathartics. Inadequate bowel preparation can result in failed detection of prevalent neoplastic lesions and has been linked to an increased risk of procedural adverse events. Previous studies have suggested that patient compliance is important to ensure proper bowel cleansing. Patient counseling along with written instructions that are simple and easy to follow and in their native language should be provided to patients.

Thus, interventions that improve the quality of bowel preparation could have a great benefit regarding colonoscopy results. Little in the literature that studies the impact of enhanced patient education on bowel preparation quality.

In this study we aim to determine the impact of patient education using telephone call one day prior to outpatient colonoscopy on bowel preparation quality.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing outpatient colonoscopy

Exclusion Criteria:

* History of previous inadequate bowel preparation
* History of colorectal surgeries
* Patient who did not sign the consent
* Patients with dementia
* Patients with Swallowing difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Bowel preparation quality | Directly after colonoscopy
  We will use Aronchick Scale as bowel preparation quality scale. This scale characterizes the percentage of the total colonic mucosal surface covered by fluid or stool, and is performed before washing or suctioning. This scale grades the adequacy of cleansing in the following:
  1. Excellent: Small volume of clear liquid, or greater than 95% of surface seen
  2. Good: Large volume of clear liquid covering 5-25% of the surface but greater than 90% of surface seen
  3. Fair: Presence of some semi-solid stool that could be suctioned or washed away but greater than 90% of surface seen
  4. Poor: Semi-solid stool that could not be suctioned or washed away and less than 90% of surface seen
  5. Inadequate: Repreparation needed Bowel preparation will be considered as adequate if the score is ≤ 3 and inadequate if the score of bowel preparation is ≥ 4.

SECONDARY OUTCOMES:
Colonic polyps rate | Directly after colonoscopy
  Detect rate of colonic polyps in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Walid Nassreddine, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon